CLINICAL TRIAL: NCT05449769
Title: Piloting a Web-based Personalised Nutrition App (eNutriCardio) With Patients Offered Cardiac Rehabilitation
Brief Title: Supporting Cardiac Rehabilitation With eNutriCardio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Royal Berkshire NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Faustina Hwang, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 301799
Record Dates: First submitted 2022-06-16; First posted 2022-07-08 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Event; Diet Habit; Diet Modification
Keywords: Food frequency questionnaire; Nutrition; Dietary intake; Diet quality; Cardiac rehabilitation; Personalised nutrition
MeSH Terms: conditions — Cardiovascular Diseases; Feeding Behavior

STUDY DESIGN:
Masking Description: Due to the nature of the study, the participants and researchers will be unblinded. Although the participants will not be explicitly told which group they are in, they will become aware of their group after completing the eNutriCardio FFQ at baseline. Those randomised to the intervention group will receive their eNutriCardio PN advice and those randomised to the control group will not receive any PN advice from eNutriCardio and therefore know which group they have been allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Those in the intervention group will receive eNutriCardio PN advice after completing the eNutriCardio FFQ at baseline only. At weeks 2, 4 and 8 of the study, participants will also receive coaching emails which includes reminders of their PN advice and questions asking them to reflect on their goal progress, if any. This will be in addition to their participation in an NHS CR programme (if they choose to join).
  Interventions: Behavioral: eNutriCardio personalised nutrition advice
- Control group (No Intervention): Those in the control group will not receive any PN advice from eNutriCardio and hence, will not receive any coaching emails. They will record their diet using eNutriCardio's FFQ . They will still be eligible to take part in an NHS CR programme.

INTERVENTIONS:
Behavioral: eNutriCardio personalised nutrition advice — eNutriCardio is a web-based app that administers an FFQ and delivers PN advice to the user. The advice is generated from their responses in the FFQ and considers their sex so the reports are unique to each participant. This report (referred to as a 'healthy eating report') will also include an interactive component, allowing the participant to reflect on the advice received and set personal healthy eating goals to motivate behaviour change. The messages presented in the report have been developed by the eNutriCardio Team, including a registered dietitian and registered nutritionist, are in line with UK dietary guidelines (primarily the EatWell Guide), and promote a Mediterranean-style diet (in line with NICE guidance). Therefore, the advice builds on the generalised advice given during the usual NHS CR programme.
  Arms: Intervention group

SUMMARY:
Following a heart attack or percutaneous coronary intervention (PCI) procedure (to 'open up' narrowed blood vessels in the heart), patients are encouraged to join a cardiac rehabilitation (CR) programme, which provides health and lifestyle advice to assist recovery and reduce risk of future cardiac events. Whilst NICE recommends that CR should "offer people an individual consultation to discuss diet", access to registered dietitians is limited. Instead, CR patients typically receive general healthy eating guidance. Since approximately 50% of patients decline CR, online tools may improve participation. The University of Reading have developed a web-based application (eNutriCardio) that uses a diet questionnaire to assess the quality ('healthiness') of a user's diet. It provides the user with unique, personalised recommendations of foods to increase/reduce to improve diet quality, which aligns with UK public health dietary advice, and incorporates behaviour change techniques.

This pilot study will investigate whether supplementing the usual NHS CR offering with personalised nutrition advice from eNutriCardio (intervention) has a different impact on diet quality and cardiac risk factors (e.g. weight and blood cholesterol) than the CR offering alone (control) after 12 weeks. 82 post-heart attack or PCI patients will provide a dried blood spot sample and record their typical diet using eNutriCardio before being randomly allocated to the control or intervention group. Both groups will be invited to participate in an NHS CR programme, but only intervention participants will receive nutrition advice from eNutriCardio. After 12 weeks, both groups will repeat the diet questionnaire and blood spot sample at home. A follow-up questionnaire will be completed after a further 8 weeks. Participants may also join an optional focus group to discuss their experiences of CR and eNutriCardio. This study is funded by the Health Innovation Partnership, a collaboration between the University of Reading and RBFT.

DETAILED DESCRIPTION:
Recruitment will end when 82 participants have been recruited or the recruitment end date (29th February 2024) is reached (whichever comes first). Participants will be screened by the experienced RBFT Cardiology Research Team following their admission to hospital for a myocardial infarction or PCI procedure. Immediately after receiving informed consent and completing the screening form, the Cardiology Research Team will direct eligible participants to eNutriCardio and help them to register. After registration, participants will be randomly allocated by eNutriCardio to either the PN intervention or control group:

* PN intervention group: in addition to the usual NHS CR offering, participants will receive web-based delivery of PN advice based on the participant's dietary intake; PN advice will be unique to each participant.
* Control group: participants will receive the usual NHS CR offering without PN advice from eNutriCardio.

Since people are often more motivated to change their diet following a 'health scare', participants will use eNutriCardio during their hospital stay or be asked to do this within 7 days of discharge to ensure their pre-event/pre-surgery diet is captured at baseline (any new 'healthier' dietary regimes would be misrepresentative of their habitual intake).

This proof-of-principle pilot study will be conducted over 20 weeks alongside the usual NHS CR offering:

* Week 0 (baseline; ideally within 7 days of hospital discharge): participants will use eNutriCardio to complete the eNutri FFQ, to provide self-reported anthropometric measurements (height and weight) and demographic information, and to answer questions on behaviour change, physical activity, computer proficiency, and usability of eNutriCardio (via the system usability scale (SUS)). They will also provide a DBS sample. Those randomised to the PN group will also receive PN advice about their diet via eNutriCardio.
* Approximately 10 days after hospital discharge: as part of the usual CR care, participants will be contacted by a CR team to discuss CR. They may choose to join or decline to take part.
* Approximately week 4-8: as part of usual CR care, participants will start their 6-8 week CR programme (unless they have declined).
* Weeks 2, 4 & 8: participants in the PN group only will receive interactive coaching emails to set goals and be reminded of their PN advice.
* Week 12 (end of study): participants in both groups will use eNutriCardio to complete the eNutri FFQ, provide self-reported weight, answer questions on physical activity and behaviour change (repeated from week 0), and provide feedback on the CR offering and dietary advice received during the study (e.g. from CR and/or eNutriCardio). They will also provide a second DBS sample.
* Week 20 follow-up: participants in both groups will complete a short online questionnaire about the longer-term effects of the dietary advice received during the study.
* Focus group: after completing the study, 8-10 participants in each group will be invited to participate in an optional focus group at the University of Reading to discuss the dietary advice in more detail.

ELIGIBILITY:
Pre-screening inclusion criteria (i.e. before patient is approached on the ward):

* Adult patients admitted to RBH following MI or elective PCI procedures
* Eligible to take part in an NHS CR programme run by RBFT or Berkshire Healthcare NHS Trust (identified as living in eligible postcode areas).

Screening inclusion criteria (i.e. screening following the consent process):

* Able to understand verbal and written English without difficulties.
* Able to access eNutriCardio from their usual location (e.g. home): will have access to a suitable device (laptop, computer, tablet or smartphone) AND access to the internet .
* Have an active email address.

Focus group inclusion criteria:

* Request to be contacted about the focus group
* Complete the eNutriCardio questionnaires during week 12
* Take part in an NHS Cardiac Rehabilitation programme
* Can visit the UoR for approximately 1 to 1½ hours
* Able and willing to contribute to a group discussion speaking in English
* Willing to be audio and video recorded
* Other inclusion criteria will already be identified through participation in the pilot study e.g. 18 years and older, able to read and understand English, do not have a dementia or another condition affecting memory

Pre-screening exclusion criteria:

* Diagnosed with dementia or other conditions affecting memory.
* Diagnosed with diabetes (any type).

Screening exclusion criteria:

* Patients unable to give informed consent.
* Pregnant, lactating or planning a pregnancy within the next 5 months.
* Food allergies to dairy, nuts/seeds and/or fish/shellfish.
* Medical conditions/treatments that have a considerable impact on an individual's diet/appetite on a day-to-day basis (e.g. severe gastrointestinal disorders, receiving chemotherapy treatment).
* Usually eat on fewer than 2 occasions per day.
* Receiving dietary advice from a dietitian, nutritionist or medical professional or plan to do so within the next 5 months.
* Following a restrictive diet, such as a vegan diet, meal replacement shake/juice diet (e.g. SlimFast), intermittent fasting diet (e.g. 5:2), very low carbohydrate diet (e.g. keto, Atkins) or any "fad"/"celebrity" diet, or plan to do so within the next 5 months; vegetarians can take part.
* Following a weight-loss programme, such as Weight Watchers, Noom, LighterLife and Slimming World, or plan to do so within the next 5 months; those aiming to lose weight through general healthy eating and "cutting down" without following specialised weight loss advice can take part.
* Taking weight-loss medication (prescribed or over the counter) or plan to do so within the next 5 months.
* Visual and/or physical impairments that prevent an individual from interacting with visual elements on the screen on their device/using their device, such as clicking buttons/mouse or using the touch pad or viewing images.
* Taking part in another research study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Diet quality score (DQS) | Baseline
  An 11-item eNutriCardio DQS will be automatically calculated by eNutriCardio after completing the FFQ. The eNutri DQS was originally developed to quantify diet quality (i.e., the healthiness of a diet) for Northern European adults and has been revised for a UK population. It is composed of 11 food and nutrient components that are summed to give an overall score, where higher scores reflect the healthiest diets based on adherence to dietary guidelines.
Diet quality score (DQS) | Week 12
  An 11-item eNutriCardio DQS will be automatically calculated by eNutriCardio after completing the FFQ. The eNutri DQS was originally developed to quantify diet quality (i.e., the healthiness of a diet) for Northern European adults and has been revised for a UK population. It is composed of 11 food and nutrient components that are summed to give an overall score, where higher scores reflect the healthiest diets based on adherence to dietary guidelines.

SECONDARY OUTCOMES:
Weight | Baseline
  Self-reported measurement of weight
Weight | Week 12
  Self-reported measurement of weight
Height | Baseline
  Self-reported measurement of height
Body mass index (BMI) | Baseline
  Automatically calculated by eNutriCardio after providing self-reported weight and height
Body mass index (BMI) | Week 12
  Automatically calculated by eNutriCardio after providing self-reported weight and height
eNutriCardio Food Frequency Questionnaire (FFQ) dietary intake data | Baseline
  eNutriCardio is a 158-item FFQ which participants will use to identify how often they typically ate/drank each item during the last 4 weeks (e.g. once a day, less than once a week, not in the last 4 weeks) then choose their typical portion size from a range of 7 photos/buttons. To increase the accuracy of the FFQ, some food/drink items have an extra question, such as the type of milk used on breakfast cereals/hot drinks or whether the food/drink item consumed was a reduced fat/sugar variety. The responses to the FFQ are used to automatically calculate the average intake in grams per day for each item.
eNutriCardio Food Frequency Questionnaire (FFQ) dietary intake data | Week 12
  eNutriCardio is a 158-item FFQ which participants will use to identify how often they typically ate/drank each item during the last 4 weeks (e.g. once a day, less than once a week, not in the last 4 weeks) then choose their typical portion size from a range of 7 photos/buttons. To increase the accuracy of the FFQ, some food/drink items have an extra question, such as the type of milk used on breakfast cereals/hot drinks or whether the food/drink item consumed was a reduced fat/sugar variety. The responses to the FFQ are used to automatically calculate the average intake in grams per day for each item.
Individual DQS component scores, food group intakes (e.g. vegetables, wholegrains) and nutrient intakes (e.g. saturated fat, sodium) | Baseline
  Recorded via eNutriCardio FFQ
Individual DQS component scores, food group intakes (e.g. vegetables, wholegrains) and nutrient intakes (e.g. saturated fat, sodium) | Week 12
  Recorded via eNutriCardio FFQ
Dried blood spot biomarkers | Baseline
  Biochemical markers of dietary intake (such as plasma fatty acids) and cardiovascular risk (such as blood total cholesterol)
Dried blood spot biomarkers | Week 12
  Biochemical markers of dietary intake (such as plasma fatty acids) and cardiovascular risk (such as blood total cholesterol)
Participants motivation and perceived ability to make dietary changes | Baseline
  Measured through a short psychology questionnaire covering ability, opportunity, motivation, and knowledge
Participants motivation and perceived ability to make dietary changes | Week 12
  Measured through a short psychology questionnaire covering ability, opportunity, motivation, and knowledge
Participant feedback on the dietary advice received from eNutriCardio and/or the NHS cardiac rehabilitation programme | Week 12
  Questionnaire covering how effective the dietary advice was at encouraging the participants to make healthy changes to their diet and whether they encountered any barriers
Participant feedback on the cardiac rehabilitation programme (or barriers preventing them from joining) | Week 12
  Questionnaire covering the type of cardiac rehabilitation programme joined (at home or in-person), if any, what their goals are for recovery and whether they would be interested in using an app that can provide advice on certain aspects of cardiac rehabilitation (e.g., diet, smoking, physical activity, weight).
Feedback on the dietary advice received (including eNutriCardio) and experience of the cardiac rehabilitation programme | Within 4 months of completing the study
  An optional focus group for participants to discuss the dietary advice they received and their experience of the cardiac rehabilitation programme. One focus group for the intervention group and one focus group for the control group.
Feedback on the longer-term impact of the dietary advice received | Week 20
  A follow-up questionnaire provided at 20 weeks after joining the study to determine whether there was a longer-term impact of the dietary advice received.
Usability of eNutriCardio measured by the System Usability Scale (SUS) | Baseline
  The SUS is a 10-item questionnaire with 5 response options that range from Strongly Agree to Strongly Disagree and is a reliable tool for measuring usability.

CONTACTS AND LOCATIONS:
Overall Officials: Faustina Hwang, Professor, Principal Investigator — University of Reading
Locations (2):
- United Kingdom (2):
  - Royal Berkshire Hospital, Reading, Berkshire
  - University of Reading, Reading, Berkshire

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymised individual participant data that underlie results in publications in a public repository. Sharing of IPD will be in line with the confidentiality and consent agreements. This may include:
  * Sociodemographics
  * Anthropometrics
  * Dietary intake data
  * Blood biomarkers
Time Frame: No later than the time of first publication and available indefinitely thereafter.
Access Criteria: We plan for open access.

REFERENCES:
- [Background] Zenun Franco R, Fallaize R, Weech M, Hwang F, Lovegrove JA. Effectiveness of Web-Based Personalized Nutrition Advice for Adults Using the eNutri Web App: Evidence From the EatWellUK Randomized Controlled Trial. J Med Internet Res. 2022 Apr 25;24(4):e29088. doi: 10.2196/29088. PMID 35468093